CLINICAL TRIAL: NCT01469624
Title: Evaluating the Protective Effect of Pentoxifylline on Contrast Induced Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, jamshid roozbeh, Clinical Professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 89-01-01-2507
Record Dates: First submitted 2011-10-25; First posted 2011-11-10 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Nephropathy
Keywords: Contrast Induced Nephropathy; Pentoxifylline; PCI
MeSH Terms: conditions — Kidney Diseases | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test group (Experimental): This group receives pentoxifylline
  Interventions: Drug: Pentoxifylline
- Control group (No Intervention)

INTERVENTIONS:
Drug: Pentoxifylline — pentoxifylline 400 mg PO three times a day for 24 hours before and 24 hours after PCI
  Other Names: Trental by Sanofi-Aventis
  Arms: Test group

SUMMARY:
Contrast induced nephropathy (CIN) is of great concern when using contrast media in the new era of medicine. CIN is defined as 25-50% relative increase, 0.5-1 absolute increase in serum creatinin value or 25% fall in GFR. The incidence of CIN is found to be 0% to 10% in general population and up to 50% in high risk population. High risk patients include those with chronic kidney disease (GFR<60 ml/min/1.73 m²) Diabetes Mellitus, congestive heart failure, anemia and advanced age. Amount and kind of contrast medium and decreased circulating blood volume are other important predictors of CIN. 50% of cases of CIN happen within 24 hours of contrast injection. Maximum creatinin levels are reached between 48-72 hours. It usually returns to previous levels in 7-10 days. Suggested mechanisms are renal vasoconstriction and tubular injury. N-acetylcysteine and hydration are proved to be protective against CIN and theophylline may have a role. In this study, it is hypothesized that pentoxifylline, a dimethylxanthine, can also protect renal cells from CIN. It has been observed that pentoxifylline improves oxygen delivery to ischemic tissues, diminishes oxidative damage to renal tissue and may also scavenge free radicals. Percutaneous coronary intervention is assumed a high risk procedure for developing CIN as the amount of contrast used in PCI is remarkable. Therefore, the patients undergoing PCI were selected for the trial. A prospective randomized trial will be conducted on patients undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

* All eligible consecutive patients who are admitted to the angiography center of university hospitals for PCI since April 2011 will be enrolled to enter the study.

Exclusion Criteria:

* Serum creatinine above 1.5 mg/dl
* Frank bleeding tendency
* Those previously on pentoxifylline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2011-04; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Serum Creatinine | 48 hours after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Jamshid Roozbeh, Nephrologist, Study Chair — Shiraz Unievrsity of Medical Sciences, Shiraz, Iran
Locations (1):
- University Hospitals, Shiraz, Fars, Iran